CLINICAL TRIAL: NCT03706378
Title: Food Modification to Alter Glycaemia and Insulinaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Collaborators: Health Promotion Board, Singapore (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017/00538
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Resistant Starch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Glucose Reference 1 (Other): 50g glucose dissolve in 250 ml of water
  Interventions: Other: Glucose Reference 1
- Glucose Reference 2 (Other): 50g glucose dissolve in 250 ml of water
  Interventions: Other: Glucose Reference 2
- Glucose Reference 3 (Other): 50g glucose dissolve in 250 ml of water
  Interventions: Other: Glucose Reference 3
- Wheat Yellow Noodle (Experimental): Boiled 170.6g of wheat yellow noodle
  Interventions: Other: Wheat Yellow Noodle
- Beta-glucan Yellow Noodle (Experimental): Boiled 230.4g of beta-glucan yellow noodle.
  Interventions: Other: Beta-glucan yellow Noodle
- Rice Roll (Experimental): Steamed 197.6g of rice roll
  Interventions: Other: Rice Roll
- Rice Roll with resistant starch (Experimental): Steamed 232.6g of rice roll fortified with resistant starch
  Interventions: Other: Rice Roll with resistant starch
- Sucrose jelly (Experimental): Jelly made with 25g of sucrose and 48g of wheat white bread
  Interventions: Other: Sucrose Jelly
- Isomaltulose jelly (Experimental): Jelly made with 25g of isomaltulose and 48g of wheat white bread
  Interventions: Other: Isomaltulose Jelly

INTERVENTIONS:
Other: Glucose Reference 1 — Glucose contains 50g of available carbohydrates
  Arms: Glucose Reference 1
Other: Glucose Reference 2 — Glucose contains 50g of available carbohydrates
  Arms: Glucose Reference 2
Other: Glucose Reference 3 — Glucose contains 50g of available carbohydrates
  Arms: Glucose Reference 3
Other: Wheat Yellow Noodle — Wheat Yellow Noodle will contain 50g of available carbohydrate
  Arms: Wheat Yellow Noodle
Other: Beta-glucan yellow Noodle — Beta-glucan yellow noodle will contain 50g of available carbohydrate
  Arms: Beta-glucan Yellow Noodle
Other: Rice Roll — Rice Roll will contain 50g of available carbohydrate
  Arms: Rice Roll
Other: Rice Roll with resistant starch — Rice Roll fortified with resistant starch will contain 50g of available carbohydrate
  Arms: Rice Roll with resistant starch
Other: Sucrose Jelly — Jelly and bread will contain 50g of available carbohydrate. The jelly will contain 25g of sucrose
  Arms: Sucrose jelly
Other: Isomaltulose Jelly — Jelly and bread will contain 50g of available carbohydrate. The jelly will contain 25g of Isomaltulose
  Arms: Isomaltulose jelly

SUMMARY:
The study specifically aims to determine glycemic and insulinemic response of added low GI ingredients, beta-glucan, resistant starch and isomaltulose to foods.

DETAILED DESCRIPTION:
There will be a total of 9 test sessions and each session will last up to 3 hours. At each test session, the following procedures will be performed: two finger-prick blood samples, five minutes apart to measure baseline blood glucose and insulin concentrations. Subject will be served the test food and to consume within15 minutes. Following the test meal, blood samples will be collected at the following time points: 15, 30, 45, 60, 90, 120, 150 and 180min for glucose measurements and insulin measurements will be collected at 30, 60, 90, 120, 150 and 180min.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males
* Chinese ethnicity
* Age ≥21 and ≤ 40 years
* Body mass index between 18.5 to 25 kg/m2
* Normal blood pressure ≤140/90 mmHg
* Fasting blood glucose <6.0 mmol/L
* In general good health

Exclusion Criteria:

* Current smoker
* Have metabolic diseases (such as diabetes, hypertension etc)
* Have glucose-6-phosphate dehydrogenase deficiency (G6PD deficiency)
* Have medical conditions and/or taking medications known to affect glycaemia (glucocorticoids, thyroid hormones, thiazide diuretics)
* Have an ongoing infection or currently undergoing treatment at the time of screening
* Have known Chronic infection or known to suffer from or have previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
* Have active Tuberculosis (TB) or currently receiving treatment for TB
* Intolerances or allergies to any foods
* Partake in sports at the competitive and/or endurance levels
* Intentionally restrict food intake

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male participants
Enrollment: 14 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Glucose | up to 180 minutes
  Blood glucose will be collected using finger prick method and analysed using Hemocue analyser
Insulin | up to 180 minutes
  Blood glucose will be collected using finger prick method and analysed using Cobas analyser

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore